CLINICAL TRIAL: NCT04769752
Title: Use and Prescription of Beta-blockers Before Cardiac Surgery With Cardiopulmopnary Bypass: Multicenter Observational Analysis of Practices and Its Association With Postoperative Morbidity-mortality.
Brief Title: Beta Blocker Use in Cardiac Surgery and Association With Postoperative Course
Acronym: BLOCK
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: Guinot 2021
Record Dates: First submitted 2021-02-23; First posted 2021-02-24 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2023-02

CONDITIONS: Cardiac Surgery With Cardiopulmonary Bypass

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- No beta-blocker: Patient do no treat with beta-blocker before the surgery
  Interventions: Other: collection of the allocated treatment; Other: collection of medical complications
- Beta blocker: Patient treat with beta-blocker in accordance to international guidelines
  Interventions: Other: collection of the allocated treatment; Other: collection of medical complications
- Beta blocker2: Patient treat with beta-blocker without respect of international guidelines

INTERVENTIONS:
Other: collection of the allocated treatment — collection of the allocated treatment
  Groups: Beta blocker; No beta-blocker
Other: collection of medical complications — collection of medical complications
  Groups: Beta blocker; No beta-blocker

SUMMARY:
The objective of this study is to describe in a cohort of cardiac surgery patients the use of beta-blockers before surgery and their maintenance or withdraw according to international recommendations in order to compare patients who receive a beta-blocker with maintenance during the surgical period (international recommendation) to those for whom prescription and maintenance are not respected. Patients are treated according to standard practice and this protocol does not change patient management. No additional information or data is required by the study other than the data usually collected in the patient record (drug treatment, medical history, operating data, postoperative data, complications, length of stay).

The objectives of this research are :

* To evaluate the proportion of patients receiving beta-blocker treatment prior to cardiac surgery.
* To evaluate the proportion of patients receiving beta-blocker treatment before cardiac surgery and complying with international recommendations for its maintenance/stop in perioperative cardiac surgery.
* To evaluate the incidence of complications and length of hospital stay in patients receiving beta-blockers based on compliance or non-compliance with recommendations.

ELIGIBILITY:
Inclusion Criteria:

* Major patient ≥ 18 years
* Patient operated cardiac surgery with cardiopulmonary bypass
* Patients who have given oral consent to participate after full information

Exclusion Criteria:

* Off pump cardiac surgery

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All consecutive cardiac surgical patients who meeet inclusion criteria with cardiopulmonary bypass
Sampling Method: Non-Probability Sample
Enrollment: 1789 (Actual)
Dates: Start 2020-06 (Actual); Primary Completion 2023-12-22 (Actual); Study Completion 2023-12-22 (Actual)

PRIMARY OUTCOMES:
Number of patients treated with beta-blocker in accordance with international guidelines | 7 days
  Number of patients treated with beta-blocker in accordance with international guidelines

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourogne, Dijon, France

REFERENCES:
- [Derived] Guinot PG, Fischer MO, Nguyen M, Berthoud V, Decros JB, Besch G, Bouhemad B. Maintenance of beta-blockers and cardiac surgery-related outcomes: a prospective propensity-matched multicentre analysis. Br J Anaesth. 2024 Aug;133(2):288-295. doi: 10.1016/j.bja.2024.04.018. Epub 2024 May 23. PMID 38789363